CLINICAL TRIAL: NCT06912243
Title: The Effect of Educational Animation on Anxiety and Fear in Children With Tympanostomy Tube Placement in Pediatric Surgery: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Aylin Kurt, Asst. Prof., Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-SBB-0907
Record Dates: First submitted 2025-03-29; First posted 2025-04-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Surgical Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational animation about the process of ear tube surgery (Experimental): A nurse will explain the process of ear tube surgery to children in an educational video. This educational video scenario includes information about a child's fears before surgery, the structure of the ear, what they are most curious about, what an ear tube is, what happens during and after surgery. The educational video will be made by a person specialized in computer technologies. Artificial intelligence will be used in the vocalization of the educational video. Expert opinion will be taken for the instructional video. The duration of the educational video is planned to be in the range of 3-4 minutes in total.
  Interventions: Other: Educational animation about the process of ear tube surgery
- Control-Standard Maintenance (Other): Children in the control group will be given the standard information given to all children who had ear tube surgery in the relevant ward.
  Interventions: Other: Control-Standard Care

INTERVENTIONS:
Other: Educational animation about the process of ear tube surgery — A nurse will explain the process of ear tube surgery to children in an educational video. This educational video scenario includes information about a child's fears before surgery, the structure of the ear, what they are most curious about, what an ear tube is, what happens during and after surgery. The educational video will be made by a person specialized in computer technologies. Artificial intelligence will be used in the vocalization of the educational video. Expert opinion will be taken for the instructional video. The duration of the educational video is planned to be in the range of 3-4 minutes in total.
  Arms: Educational animation about the process of ear tube surgery
Other: Control-Standard Care — The standard information given to all children who had ear tube surgery in the relevant ward will be given to the children in the control group.
  Arms: Control-Standard Maintenance

SUMMARY:
The study was planned as a randomized controlled experimental research to determine the effect of educational video screening on anxiety and fear in children. All children between the ages of 6-10 years old who underwent ear tube surgery will be included. Children will be randomly assigned to two groups (training video group, control group-standard care). In the training video group, a nurse will explain the process of ear tube surgery to the children with an educational video. The scenario of this educational animation will include information about the preoperative fears of a child who will undergo ear tube surgery, the structure of the ear, what they are most curious about, what the ear tube is, what will happen during and after surgery. In the control-standard care group, the standard information given to all children who had ear tube surgery in the relevant service will be given to the children in the control group. Data will be collected with the Sociodemographic Questionnaire, Child Anxiety Scale-Condition Child Fear Scale before and after surgery.

DETAILED DESCRIPTION:
When a child becomes ill and undergoes surgery, it can be an event that increases anxiety and fear for both the child and the parents. Parents may experience significant decision conflicts when making decisions about their child's elective surgical treatment, such as ear tube surgery. Children encounter many situations in the hospital that cause anxiety and fear. Especially if there is a surgical intervention plan in the treatment plan of the disease, psychological problems may arise in the child and family members. During the preoperative period, children can be quite stressed. Anxiety-inducing conditions include feeling restless due to the operation, fear of loneliness, feeling of foreignness, fear of pain after surgery, concern about disruption of the integrity of the body and frequent use of medical terms. Reducing anxiety before surgery has positive results in the recovery of the sick child and the parent after surgery. Methods such as preanesthetic drugs, distractions, the presence of the parent with the patient before anesthesia, preoperative training and psychological preparation of both the child and the family for surgery are used to reduce preoperative anxiety.

In the study examining the content of social media posts about ear tubes in children on popular social media platforms Instagram and Facebook, it was determined that most of the posts were made by parents/caregivers in the perioperative period and the rate of educational posts was low. With the increasing importance of patient/family-centered participation in the decision-making process in healthcare services, standardizing the content and increasing the usability of educational materials for surgical procedures commonly performed in children such as ear tube placement should be a priority. Since there are no standardized guidelines on how to write online patient education materials, online patient education materials vary in quality and readability.

This study may provide important information about the ear tube surgery procedure by helping children to focus their attention on positive things rather than stressful events with video and musical interventions, which are both economical and easy to use. To the best of our knowledge, there is no study in the literature examining the effect of video screening on anxiety and fear in children undergoing ear tube surgery. Therefore, this randomized controlled trial was planned to determine the effect of educational video screening on anxiety and fear in children.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-10 years old
* Having ear tube surgery
* Signing the informed consent form by the patient's legal guardian

Exclusion Criteria:

* Previous surgical operation of the child
* The child has had a cleft palate or lip operation before
* Conditions that may prevent communication with parents (e.g. language problem)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
The mean score of the Children's Anxiety Scale-Situation of the children who watched educational videos after the educaiton video was lower than that of the control group. | 12 months
  The mean score of the Children's Anxiety Scale-Situation of the children who watched educational videos after the educaiton video was lower than that of the control group.
The mean score of the Children's Fear Scale of the children who watched educational videos after the education video was lower than that of the control group. | 12 months
  The mean score of the Children's Fear Scale of the children who watched educational videos after the education video was lower than that of the control group.

SECONDARY OUTCOMES:
Children who watched educational videos had lower mean scores on the Child Anxiety Scale-Situation after the educational video compared to before the educational video. | 12 months
  Children who watched educational videos had lower mean scores on the Child Anxiety Scale-Situation after the educational video compared to before the educational video.
Children who watched educational videos had lower mean scores on the Child Fear Scale after the educational video compared to before. | 12 months
  Children who watched educational videos had lower mean scores on the Child Fear Scale after the educational video compared to before.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Merkez, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No